CLINICAL TRIAL: NCT06617702
Title: ASPIRE to Change: Leveraging Text Messaging Peer Support Coaching to Mitigate Hazardous Alcohol Consumption in Non-Collegiate Young Adults
Brief Title: Accountability Support Through Peer-Inspired Relationships and Engagement (ASPIRE) Trial
Acronym: ASPIRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Brian Suffoletto, Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 76956; 1R01AA030986-01A1 (NIH)
Record Dates: First submitted 2024-09-26; First posted 2024-09-27 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Alcohol Consumption
Keywords: alcohol; text message; young adults; peers
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A text message alcohol intervention focused on cognitive, behavioral, and peer influences (Experimental)
  Interventions: Behavioral: A text message alcohol intervention focused on cognitive, behavioral, and peer influences
- A text message alcohol intervention focused on cognitive and behavioral influences (Active Comparator)
  Interventions: Behavioral: A text message alcohol intervention focused on cognitive and behavioral influences

INTERVENTIONS:
Behavioral: A text message alcohol intervention focused on cognitive, behavioral, and peer influences — Each Thursday and Sunday ASPIRE will conduct brief text message communication aimed at modifying cognitive (e.g.desire to get drunk), behavioral (e.g.alcohol consumption), and peer influences (e.g.peer pressure and support).
  Arms: A text message alcohol intervention focused on cognitive, behavioral, and peer influences
Behavioral: A text message alcohol intervention focused on cognitive and behavioral influences — Each Thursday and Sunday ASPIRE will conduct brief text message communication aimed at modifying cognitive (e.g. desire to get drunk) and behavioral (e.g. alcohol consumption) influences.
  Arms: A text message alcohol intervention focused on cognitive and behavioral influences

SUMMARY:
This project aims to test the efficacy of a text message intervention, ASPIRE, designed to address cognitive and behavioral elements and modify exposure to peers that influence drinking behaviors. Young adults who are contemplating reducing their drinking will be recruited from a national sample and randomized to ASPIRE versus a text message intervention focused solely on cognitive and behavioral elements. We will measure effectiveness at 3, 6, and 12 months, study mechanisms driving behavior change, and identify which subgroups stand to benefit most.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-25 years (verified using date of birth)
* Lives in the U.S. (based on zip code)
* English reader (verified based on completing screen)
* 2+ days with ≧4 standard alcohol drinks for women or ≧5 standard alcohol drinks for men in past month
* Owns a mobile phone with SMS (verified by texting enrollment procedure)

Exclusion Criteria:

* Currently enrolled or past enrollment in a 4-year college
* Active military
* Pregnant or pregnancy plans in the next 12-months
* Prisoner status
* Current or planned treatment for alcohol or substance use disorder in next 12-months

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of Binge Drinking Days (BDD) | 3, 6, and 12 months
  We define BDD as a day when a woman reports 4 or more standard drinks or a man reports 5 or more standard drinks, as this equates to the alcohol consumption that raises blood alcohol concentration to 0.08 g/dl or above.

SECONDARY OUTCOMES:
Negative Alcohol Consequences (NAC) Scale Score | 3, 6 and 12 months
  We calculate the number of NAC using the Brief Young Adult Alcohol Consequences Questionnaire (B-YAACQ). The B-YAACQ is a 24-item measure of alcohol-related problems that utilizes a dichotomous (present or absent) scoring format. Higher scores indicate both wider variety and more severe pattern of alcohol-related problems.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Suffoletto, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All test message and web-based data from baseline through 12-month followups will be uploaded to the data repository (the National Institute on Alcohol Abuse and Alcoholism Data Archive (NIAAADA).
Supporting Information: Study Protocol
Time Frame: Data will be available within 1 year of study completion and available indefinitely.
Access Criteria: Individuals can request access to study data through the NIAAADA. If there are data from the trial not submitted to the NIAAADA , investigators can submit an abstract of their research question to the PI and study investigators for review. The written data request abstract will include the researcher's resume and qualifications (including a statement of any conflicts of interest), an outline of the analysis aims, analysis methods, variables requested, data to be analyzed, proposed product of the request (e.g., conference presentation, manuscript) and timeline for completion. The PIs and study investigators will review the data request abstract, and approve or decline the data request. Individuals whose data request is approved are asked to sign a confidentiality and data sharing agreement prior to receipt of any study data. The investigator making the request must obtain approval from their institution's IRB to conduct the proposed analyses.

REFERENCES:
- [Background] Kahler CW, Hustad J, Barnett NP, Strong DR, Borsari B. Validation of the 30-day version of the Brief Young Adult Alcohol Consequences Questionnaire for use in longitudinal studies. J Stud Alcohol Drugs. 2008 Jul;69(4):611-5. doi: 10.15288/jsad.2008.69.611. PMID 18612578
- [Background] Sobell LC, Brown J, Leo GI, Sobell MB. The reliability of the Alcohol Timeline Followback when administered by telephone and by computer. Drug Alcohol Depend. 1996 Sep;42(1):49-54. doi: 10.1016/0376-8716(96)01263-x. PMID 8889403
- [Background] Rueger SY, Trela CJ, Palmeri M, King AC. Self-administered web-based timeline followback procedure for drinking and smoking behaviors in young adults. J Stud Alcohol Drugs. 2012 Sep;73(5):829-33. doi: 10.15288/jsad.2012.73.829. PMID 22846247